CLINICAL TRIAL: NCT01004536
Title: A Randomized Investigator-blind Multi-center Prospective Study for the Efficacy and Safety of Silicon Gel (Dermatix) in the Prevention of Hypertrophic Scar in Subjects Undergoing Caesarean Section
Brief Title: An Investigator-blind Multi-center Prospective Study for the Efficacy and Safety of Silicon Gel (Dermatix)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Kyunghee University Medical Center (Other); Inovail (Unknown)
Responsible Party: Joo-Heung Lee, MD/professor and chair of dermatology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-08-092
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Hypertrophic Cicatrix
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- no treatment (No Intervention): The other half of cesarean section wound that is to be left untreated.
  Interventions: Other: no treatment
- silicone gel (Experimental): Randomly-designated half of cesarean section wound that is to be subject to application ot silicone gel
  Interventions: Device: silicone gel

INTERVENTIONS:
Device: silicone gel — twice daily application onto designated half of cesarean section wound for 12 weeks
  Other Names: Dermatix
  Arms: silicone gel
Other: no treatment — left untreated during the study period
  Arms: no treatment

SUMMARY:
Silicone gel is a self-drying silicone polymer that forms thin film after application onto the skin. Because silicone film is a medical device, silicone gel is also regarded as a medical device. Silicone gel has been on the market for many years for the management of scar in the phase of treatment as well as in the phase of prevention. In contrast to other methods that are expensive, invasive or inconvenient, silicone gel is convenient, non-invasive and also reasonably priced. However, the number of well-designed clinicial trials for efficacy and safety are not enough to provide robust evidences in making clinical decisions for scar management options. In a prospective, multi-center, investigator-blind randomized half-split study for patients undergoing cesarean sections, the investigators attempt to provide valid information for the efficacy and safety of silicone gel in the prevention phase of scar.

DETAILED DESCRIPTION:
Prospective subjects will be enrolled in the trial when eligibility screening and informed consent were made. One day after stitch out for cesarean sections, subjects will be asked to start applying silicone gel as the instruction to the randomly designated half of the wound 2 times a day for 12 weeks. Subjects are asked to make visits on week 4, 8, and 12 for efficacy, safety and compliance evaluations. Obstetricians, dermatologists and medical imaging specialists are involved in the trial for the evaluation of efficacy, safety and compliance. Sample size calculation as well as statistical analysis will be conducted by a designated statistician. Study product will be provided by the manufacturer at no cost and patient visits and relevant lab exams will be conducted free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female of 20-45 in ages equal to or beyond 34th of pregnancy
* Those who understand and agree on the trial conditions

Exclusion Criteria:

* Keloid (by present and past medical history)
* Secondary infection, and/or dermatitis in and around c/s wound
* Hypersensitivity to the study agent
* Diabetes
* (Pre)eclampsia

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
summation of scar scores of modified Vancouver Scar Scale | week 12

SECONDARY OUTCOMES:
summation of scar scores of mVSS 4 and 8 weeks after application | weeks 4, 8, 12
scar thickness 12 weeks after application | weeks 4, 8, 12
subjective satisfaction 12 weeks after application (VAS) | weeks 4, 8, 12
tolerability 4, 8, 12 weeks after application (index3) | weeks 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Heung Lee, MD, Study Chair — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Seoul, Seoul
  - Kyung-Hee University Medical Center, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul